CLINICAL TRIAL: NCT02170883
Title: EmPhAsIS: Empowering Pharmacists in Asthma Management Through Interactive SMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: WelTel (Unknown); College of Pharmacists of British Columbia (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Mary De Vera, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H14-01451
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Asthma
Keywords: asthma; mHealth; cluster randomized controlled trial; pharmacy practice; pharmacist
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive SMS (Experimental): Intervention with interactive SMS (text messaging) by which patients are asked to disclose their level of agreement with the following statement "I follow my asthma medication plan" and pharmacist follow-up
  Interventions: Other: Interactive SMS
- Usual care (Active Comparator): Pharmacist conducted patient education, counseling and action-plan
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Interactive SMS
  Arms: Interactive SMS
Other: Usual care
  Arms: Usual care

SUMMARY:
Between 8% and 12% of Canadians suffer from asthma. Although there are effective and inexpensive treatments, adherence to asthma treatment is amongst the lowest for all chronic diseases.The purpose of this study is to determine whether enhancing the role of community pharmacists in asthma management using interactive short messaging service (SMS) with asthma patients is a cost-effective model that will improve adherence to inhaled corticosteroid medications compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* individuals who fill a (incident or prevalent) prescription for inhaled corticosteroids (either monotherapy or in combination inhaler with long-acting beta-agonists) who have been diagnosed by a doctor as having asthma
* possessing a cell-phone with ability to send/receive text messages
* residing in British Columbia (BC), Canada and planning to reside in BC for the next 12 months
* registered with the medical services plan (MSP, the provincial insure of medically-required services) in the past 12 months, and planning to remain registered for the next 12 months
* designated pharmacy being the main drugstore for patient
* not participating in another interventional study
* consent to participate in the study.

Exclusion Criteria:

* Unable to communicate in English
* Under 14 years of age

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2015-05; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Adherence to inhaled corticosteroid medication | 12 months
  Adherence assessed by medication possession ratio

SECONDARY OUTCOMES:
Asthma control | Baseline
  Asthma control assessed by the Asthma Control Test
Asthma control | 6 months
  Asthma control assessed by the Asthma Control Test
Asthma control | 12 months
  Asthma control assessed by the Asthma Control Test
Quality of life measured by the Asthma Quality of Life Questionnaire | Baseline
  Quality of life measured by the Asthma Quality of Life Questionnaire
Quality of life measured by the Asthma Quality of Life Questionnaire | 3 months
  Quality of life measured by the Asthma Quality of Life Questionnaire
Quality of life measured by the Asthma Quality of Life Questionnaire | 12 months
  Quality of life measured by the Asthma Quality of Life Questionnaire
Health care resource utilization | 12 months
  Asthma-related hospital admissions and emergency department visits
Use of reliever medication for acute asthma attacks | 12 months
  Use of reliever medication for acute asthma attacks

CONTACTS AND LOCATIONS:
Overall Officials: Mary De Vera, PhD, Principal Investigator — University of British Columbia
Locations (1):
- UBC, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] De Vera MA, Sadatsafavi M, Tsao NW, Lynd LD, Lester R, Gastonguay L, Galo J, FitzGerald JM, Brasher P, Marra CA. Empowering pharmacists in asthma management through interactive SMS (EmPhAsIS): study protocol for a randomized controlled trial. Trials. 2014 Dec 13;15:488. doi: 10.1186/1745-6215-15-488. PMID 25494702